CLINICAL TRIAL: NCT00204347
Title: Effective Measurement of Risperidone Treatment Outcome for Persons With Borderline Personality Disorder: The UAB Borderline Rating Scale (BRS)
Brief Title: Effective Measurement of Risperidone Treatment Outcome for Persons With Borderline Personality Disorder
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Alabama at Birmingham (Other)
Collaborators: Janssen Pharmaceutica (Industry)
Responsible Party: Principal Investigator, Roberta May, Associate Professor, University of Alabama at Birmingham
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RIS-DED-WTJ
Record Dates: First submitted 2005-09-13; First posted 2005-09-20 (Estimated); Last update posted 2021-06-10 (Actual); Status verified 2021-06

CONDITIONS: Borderline Personality Disorder
Keywords: risperidone
MeSH Terms: conditions — Borderline Personality Disorder | interventions — Risperidone

INTERVENTIONS:
Drug: risperidone

SUMMARY:
The objective of Study A is to evaluate the efficacy of risperidone on the 4 behavioral dimensions of Berderline Personality Disorder (BPD)in an open label trial:mood swings, impulsivity, thing difficulties and disturbed relationships. The secondary objective of this study (Study B)is to validate a self-report measure of clinical symptoms specific to the treatment of patients with BPD, the UAB Borderline Rating Scale(BRS).

DETAILED DESCRIPTION:
Study A: An open-label, prospective trial of the efficacy and safety of risperidone in the treatment of BPD.The study is 8 weeks in duration, with a screening visit and follow-up visits at the end of Weeks 1,2,3,4,6, and 8. 20 female patients, 19 years or older will be recruited. A full medical and psychiatric history will be taken and a physical exam will be performed by a sstudy physician. A psychosocial assessment will be conducted during the screen.

Study B: The ofjective is to validate the UAB BRS by administering the BRS and other neuropsychological instruments as repeated measures over a 6 week period to 40 patients with BPD.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of BPD

Exclusion Criteria:

* Any other Axis I diagnosis except dysthymia, PTSD, or generalized anxiety disorder;substance abuse within a month; unstable medical illness.

Min Age: 19 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20
Dates: Start 2003-07; Primary Completion 2007-10 (Actual); Study Completion 2007-10 (Actual)

PRIMARY OUTCOMES:
Clinical Global Impression
Brief Symptom Inventory

SECONDARY OUTCOMES:
Beck Depression Inventory
Quality of Life Enjoyment and Satisfaction Questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Celia T. Huston, PhD, Principal Investigator — University of Alabama at Birmingham
Locations (1):
- University of Alabama at Birmingham, Birmingham, Alabama, United States